CLINICAL TRIAL: NCT01570049
Title: A Multicenter, Single Arm Clinical Trial in Patients With Rituximab Refractory B-cell Indolent Lymphoma
Brief Title: Safety and Efficacy Study of Bendamustine to Treat Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Lanjin Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGB-NHL
Record Dates: First submitted 2012-03-29; First posted 2012-04-04 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Non-Hodgkin Lymphoma by Clinical Course
Keywords: Single arm; Open label; Bendamustine HCl; Non-hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bendamustine (Experimental): Dose of 120 mg/m2/day on Day 1 and Day 2 of each treatment cycle (every 21 days), to a maximum of 8 cycles.
  Interventions: Drug: Bendamustine

INTERVENTIONS:
Drug: Bendamustine — for injection

SUMMARY:
The purpose of this study is to determine whether bendamustine HCl for injection is safe and effective in the treatment of Rituximab refractory or relapsed B-cell indolent lymphoma.

DETAILED DESCRIPTION:
This is multicenter, open label study to evaluate the safety and efficacy of bendamustine HCl in patients with indolent Non-hodgkin's lymphoma and relapsed after rituximab treatment. This injection will be given through i.v. infusion in >= 60 minutes on days 1 and 2 of every 21-day treatment cycle. Patients will be treated for up to 8 cycles unless progressive disease or unacceptable toxicity take place. Patients will be followed for up to 1 year before evaluating progression free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years
* B-cell indolent lymphoma proved by biopsy, exclude CLL/SLL
* Rituximab refractory or relapsed lymphoma patients
* At least 1 measurable tumor with shortest diameter being of > 1.0cm and longest diameter being of > 1.5cm
* ECOG PS ≤ 2
* Anticipated Survival is more than 3 months
* Hematopoietic function is normal during 14 days before enrollment (unless those abnormities related to lymphoma aggression), including: hemoglobin (Hb) ≥ 8.0g/dl (5.0mmol/L); absolute neutrophil count (ANC) ≥ 1.5X109/L; Platelet count (PLT) ≥ 80X109/L. Acceptable range for abnormities related to lymphoma aggression: Platelet count (PLT) ≥ 50X109/L; White blood cell count (WBC) ≥ 3.5X109/L; Absolute neutrophil count (ANC) ≥ 1.0X109/L
* Female subjects should not be pregnant and breast-feed, should have contraceptive method during the clinical trial and 12 months thereafter.
* Subject (or his/her legal representative) agrees to participate the trial and sign the informed consent form

Exclusion Criteria:

* Those who can not tolerate bendamustine treatment according to investigators view
* Transferred to high grade malignant lymphoma (from low grade follicular lymphoma)
* 3b grade follicular lymphoma
* With central nervous system diseases or medical history (e.g., central nervous system lymphoma or lymphoma related meningitis )
* With other anticancer treatment during the last 4 weeks
* Regularly administrated corticosteroid during the last 4 weeks, unless the dose is less or equivalent to 20mg/d prednisone
* Had tumors or have other tumors, not including non-melanoma skin cancers and cervical carcinoma in situ be treated properly
* Underwent surgical operation within 28 days before enrollment (exclude lymph node biopsy)
* Renal disfunction: serum creatinine is more than 1.5 times of upper limit of normal value
* Hepatic insufficiency: serum total bilirubin is > 1.5 times of upper limit of normal value; AST, ALT is > 2.5 times of upper limit of normal value
* Known HIV infection or HBV, HCV related active infections; HBsAg is positive; HBcAb is positive and virus copy number is > 1000
* For patients with other severe medical diseases interfering with their participations of this study(e.g., infections and diabetes not controlled well, gastric ulcer, other lung diseases, active autoimmune diseases), the suitability of participation is judged by investigators
* Patients participated in other clinical studies and got medical treatments within 30 days prior to enrollment of this trial
* Other medical and psychological conditions that influence the patients participation or signing of informed consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR=CR+PR) of bendamustine hydrochloride in patients who are refractory to rituximab therapy. | 18 months

SECONDARY OUTCOMES:
Safety profile of Bendamustine hydrochloride in this patient population | 18 months
Progression free survival (PFS) | 18 months
Overall survival (OS) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Huaqing Wang, master, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China